CLINICAL TRIAL: NCT00727493
Title: Evaluation of the Influence of Alendronate on Wound Healing After Dental Implants in Patients With Osteoporosis
Brief Title: Osteoporosis and Dental Implant
Acronym: OPOZAHN
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Prof. Dr. med. Dieter Felsenberg, Center for Muscle and Bone Research
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OPOZAHN
Record Dates: First submitted 2008-07-31; First posted 2008-08-04 (Estimated); Last update posted 2008-08-04 (Estimated); Status verified 2008-08

CONDITIONS: Osteoporosis
Keywords: osteoporosis,; bisphosphonate; therapy; dental implant
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): alendronate once weekly 70mg, calcium 1000mg and Vitamin D 800 IU daily, dental implant
  Interventions: Drug: alendronate once weekly 70mg
- 2 (Placebo Comparator): placebo once weekly, calcium 1000mg and Vitamin D 800 IU daily; dental implant
  Interventions: Drug: placebo
- 3 (No Intervention): dental implant, calcium 1000mg and Vitamin D 800 IU daily

INTERVENTIONS:
Drug: alendronate once weekly 70mg — alendronate once weekly 70mg, calcium 1000mg and Vitamin D 800 IU daily for 12 months, dental implant
  Arms: 1
Drug: placebo — placebo once weekly; calcium 1000mg and Vitamin D 800 IU daily, dental implant
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the influence of alendronate therapy on the wound healing after dental implants in patients with osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women > 2 years after menopause
* Age between 60 and 75 years
* Possibility to insert a dental implant
* Osteoporosis as defined by WHO criteria (intervention group), or women without osteoporosis / osteopenia (non-intervention group)

Exclusion Criteria:

* Pathological findings in the jaw bone
* Chronic inflammatory rheumatoid disease
* Bisphosphonate treatments during the last 12 months
* Inflammatory or metabolic bone disease, excluding osteoporosis
* Systemic corticosteroid treatments of more than one month within previous 12 months
* Severe diseases with life expectancy less than one year or expectation of rapid worsening within one year

Ages: 60 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2004-01; Primary Completion 2010-01 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
Dental CT | baseline, and 3,6,12 months after baseline

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Felsenberg, Prof. D.r, Study Chair — Leader of the center for muscle and bone research, Charité
Locations (1):
- Centre for Muscle and Bone Research, Charité - Campus Benjamin Franklin, Berlin, Germany